CLINICAL TRIAL: NCT05799651
Title: A Randomised, Double-Blind, Dose-Escalation Phase I Study in Healthy Adults to Assess the Safety, Tolerability and Immunogenicity of Glycovax-002, a Novel Vaccine Candidate Against COVID-19
Brief Title: Safety and Immunogenicity of Glycovax-002 Vaccine in Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Glycovax Pharma Inc. (Industry)
Collaborators: Government of Canada (Other Government); JSS Medical Research Inc. (Industry); Avance Clinical Pty Ltd. (Industry); Seppic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GLY-GVX-002-001
Record Dates: First submitted 2023-03-10; First posted 2023-04-05 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: SARS-CoV-2
Keywords: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Step 1 (Low Dose) (Experimental): A total of 12 participants will receive three injections, spaced by two weeks, of Glycovax-002 Low Dose or placebo (ratio 3:1).
  Interventions: Biological: Glycovax-002
- Step 2 (Medium Dose) (Experimental): A total of 12 participants will receive three injections, spaced by two weeks, of Glycovax-002 Medium Dose or placebo (ratio 3:1).
  Interventions: Biological: Glycovax-002
- Step 3 (High Dose) (Experimental): A total of 12 participants will receive three injections, spaced by two weeks, of Glycovax-002 High Dose or placebo (ratio 3:1).
  Interventions: Biological: Glycovax-002

INTERVENTIONS:
Biological: Glycovax-002 — Intramuscular injection of vaccine against SARS-CoV-2

SUMMARY:
Glycovax Pharma has developed a glycoconjugate vaccine candidate called Glycovax-002 to fight the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at the origin of COVID-19.

The aim of the study is to assess the safety, reactogenicity and immunogenicity of Glycovax-002 in humans. The study is a phase I, placebo-controlled, dose-escalation study conducted in 36 healthy females and males aged between 18 and 55 years old. The vaccine will be administered three times with a two-week time interval between each dose.

Dose escalation is conducted in three steps. At each step, 9 participants receiving the vaccine will be randomized with 3 participants receiving placebo (normal saline). Progression to next step is conditional to a DSMB's approval.

ELIGIBILITY:
Inclusion Criteria:

All the following criteria need to be met for inclusion:

1. Adults in good health as determined by the Principal Investigator or Sub-Investigator between 18 - 55 years old inclusively.
2. Able to provide informed consent and willing to comply with the study procedures.
3. BMI ≥ 18.0 kg/m2 and ≤ 35.0 kg/m2, with weight ≥ 45 kg for female subjects and ≥ 50 kg for male subjects.
4. Vital signs within the following limits: systolic blood pressure (BP) 90 - 140 mmHg, inclusive; diastolic BP 40 - 90 mmHg, inclusive; heart rate 40 - 100 bpm, inclusive; respiratory rate 10 - 22 bpm, inclusive; temperature 35.5 - 37.5 °C, inclusive.
5. Women of child-bearing potential should have a negative serum pregnancy test at Screening and a confirmatory negative urine pregnancy test at Baseline (Day 0, defined as enrolment), one before the second administration (Day 14) and one before the third and last dose administration (Day 28).
6. Agrees to practice acceptable contraception during the study if female of child-bearing potential or male partner of female of child-bearing potential.
7. Physical examination, clinical assessments, and laboratory values within normal limits during Screening, unless assessed as not clinically significant by Investigator or Delegate.
8. Has received a dose or multiple doses, of a registered COVID-19 vaccine, with the last dose more than two months prior to enrolment.

Exclusion criteria:

Participants will be excluded if any of the following criteria are met:

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator, that could adversely affect the safety of the participant or confound the results of the study. Fully resolved childhood asthma is not exclusionary.
2. History of malignancy, except for non-melanoma skin cancer when excised more than two years ago and cervical intraepithelial neoplasia that has been successfully cured more than two years prior to Screening.
3. Any of the following specific conditions:

   1. Autoimmune conditions;
   2. Metabolic disorders;
   3. Glycosyl transferase disorders (including disorders of fucosyl transferase and fucose metabolism);
   4. Tn polyagglutination of erythrocyte syndrome, deficiency of galactosyl transferase, anemia, leukopenia, or thrombocytopenia;
   5. Known bacterial infections involving neuraminidase-expressing bacteria.
4. Use of any prescription medication that, in the Investigator's judgment, can interfere with the interpretation of the study tests or in the opinion of the Investigator may be contra-indicated for use with Glycovax-002. Medications that have been stable in the past 3 months may be allowed, for instance medications for hypertension, hypercholesterolemia, and gastroesophageal reflux disease (e.g. proton pump inhibitors).
5. Receipt of chronic systemic treatment with known immunosuppressant medications, or radiotherapy, within 60 days prior to enrolment.
6. Receipt of chronic systemic immunostimulant therapy (such as interferons or interleukins) within 60 days prior to enrolment.
7. Receipt of systemic corticosteroids (≥20 mg/day of prednisone or equivalent) for ≥14 days within 28 days prior to enrolment.
8. Receipt of blood/plasma products or immunoglobulins within 6 months prior to enrolment.
9. Receipt of any anticoagulation treatment (other than low dose aspirin).
10. History of myocarditis or pericarditis.
11. Presence of any sign or symptom that may suggest an active respiratory infection including COVID-19 at enrolment.
12. Any vaccination other than for influenza within 60 days prior to enrolment, or an influenza vaccination within 30 days prior to enrolment.
13. Planning to receive vaccination within 60 days after enrolment in the study.
14. Positive testing for COVID-19 within 3 months of enrolment or positive PCR testing for COVID-19 at enrolment.
15. Diagnosed with Influenza within 30 days prior to enrolment.
16. Positive for infection with HIV or with hepatitis B or C at Screening.
17. Receipt of an investigational drug within 30 days or 5 half-lives (whichever is longer) before study enrolment. For studies involving investigational products that fall within the categories mentioned in other Inclusion Criteria, the respective timelines should be respected.
18. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g., anaphylaxis).
19. History of hypersensitivity or allergic reaction to any of the components of GVX-002, including diphtheria toxoid, or squalene-based adjuvants, including Sepivac SWE™ and MF59.
20. History of drug or alcohol abuse, or positive detection test at Screening or prior to Study Drug administration for alcohol or any illicit drug including cannabis.
21. Current smoking (more than 10 cigarettes/week), current vaping (more than 80 puffs/week), current cannabis use, alcohol abuse (defined as regularly consuming more than 14 units of alcohol per week), or current drug abuse (as tested at Screening), to avoid possible impairment of immune function.
22. Presence of tattoos or scars on the upper arms that would preclude visualising any injection site reactions.
23. Any other reason (e.g., poor venous access) at the Investigator's discretion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the overall safety and reactogenicity of the Glycovax-002 conjugated vaccine administered at three different doses in healthy adults. | Day 0 - 360
  Safety:
  * Incidence of Adverse Events (AEs) in all participants.
    * Occurrence of each solicited local and systemic AE, during each 7-day follow-up period after injection.
    * Occurrence of any AEs until 28 days after the last injection.
    * Occurrence of serious AEs until one year after the first injection.
  * Assessment of safety will involve blood tests for biochemistry, hematology, serum chemistry and immunogenicity, urine tests for urinalysis, and participant diaries.
  Reactogenicity:
  Reactogenicity will be assessed by the incidence of the following solicited reactions for the first 7 days after each administration:
  Local:
  * Swelling at injection site
  * Erythema at injection site
  * Pain at injection site
  General (systemic):
  * Fever
  * Fatigue
  * Chills
  * Diarrhea
  * Myalgia
  * Arthralgia
  * Headache
  * Nausea/Vomiting

SECONDARY OUTCOMES:
To assess the immunogenicity induced by Glycovax-002 in healthy adults | Day 0 - 120
  Immunogenicity will be assessed prior to each dose of Glycovax-002 and then at 1 and 3 months after the last dose, i.e. at Days 0, 14, 28, 56 and 120, except otherwise stated.
  * Serum anti-TF IgG
  * Total serum IgG, IgA, and IgM
  * Cytokine (Th1 and Th2) concentration in serum, at baseline and six hours after the last Glycovax-002 administration on Day 28:
    * IFN-γ
    * TNF-α
    * IL-2
    * IL-4
    * IL-13
  * CD4 and CD8 T-cell and B-cell counts and CD4/CD8 ratio.
To assess the virus-neutralizing antibody response induced by Glycovax-002 in healthy adults | Day 0 - 56
  SARS-CoV-2 virus-neutralising antibody levels in serum, on Days 0 and 56 only, by a pseudovirus neutralisation assay
  * based on the original Wuhan viral strain, and
  * based on the latest Variant of Concern available for testing at time of study initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Kristi McLendon, MD, Principal Investigator — Nucleus Network
Locations (1):
- Q-Pharm Pty Ltd, Herston, Queensland, Australia